CLINICAL TRIAL: NCT07138924
Title: Comparative Analysis Of Graston Technique Versus Dynamic Oscillation Stretching Technique For High Heel Users And Its Impact On Body Posture
Brief Title: Graston Technique vs Dynamic Oscillation Stretching Technique For High Heel Users And Its Impact On Body Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/02012
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hyperlordosis
Keywords: Hyperlordosis Anterior pelvic tilt Graston Technique Dynamic Oscillating Stretch
MeSH Terms: conditions — Swayback

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graston Technique (Experimental): Experimental Group A: Graston technique on calf and Paraspinal (erector spinae) muscles with conservative physiotherapy treatment plan i.e. hot pack for 10-15 min (calf muscles) calf stretches (10 reps x 2 sets) and post session cold pack for 5 min.
  Interventions: Other: Graston Technique
- Dynamic Oscillatory Stretch Technique (DOST) (Active Comparator): Experimental Group B: Dynamic oscillation stretching technique on gastrocnemius, soleus, and hamstring with conservative physiotherapy treatment plan i.e. hot pack for 10-15 min (calf muscles) calf stretches (10 reps x 2 sets) and post session cold pack for 5 min.
  Interventions: Other: Dynamic Oscillatory Stretch Technique

INTERVENTIONS:
Other: Graston Technique — Firstly, apply a moisturizer or gel to affected part. Then gentle strokes are applied from proximal to distal direction to assess trigger point or taut band. After knowing the exact area, apply strokes gently with minimum force in all directions by keeping tool in 30- 60-degree angle. Total Application time will be between 40-120 seconds. conservative physiotherapy treatment plan is hot pack for 10-15 min, calf stetches 10 reps x 2 sets and post session cold pack for 5 min. Home exercise plan is william training i.e. single knee to chest, double knee to chest, pelvic tilts, iliospoas stretch, hamstring stretch and squat (10reps x1 set)
  Arms: Graston Technique
Other: Dynamic Oscillatory Stretch Technique — Passively stretch that is at the first point of stretch sensation. The next component to DOS, 2-sec, passive stretch with slow oscillation. Total 10 reps x 2 sec hold oscillations x 3 sets.conservative physiotherapy treatment plan is hot pack for 10-15 min, calf stetches 10 reps x 2 sets and post session cold pack for 5 min. Home exercise plan is william training i.e. single knee to chest, double knee to chest, pelvic tilts, iliospoas stretch, hamstring stretch and squat (10reps x1 set)
  Arms: Dynamic Oscillatory Stretch Technique (DOST)

SUMMARY:
In high heel users, most of the previous work has focused on the lower limb. However, we did not find any study that specifically targeted the lumbar region. The novelty of this study lies in raising awareness that high heel users experience a full-body postural disturbance. While studies had involved the lower limb, but it is crucial to also include the lumbar region. This is because high heel users often feel more pain in the lower limb, which may be leading us to focus solely on lower limb and neglect the lumbar region. However, the mechanics of the lumbar region are also deteriorating along with the lower limb, which may lead to musculoskeletal related issues to high heel users in future. In Pakistan, no previous research is conducted, That compare the effect of Graston Technique Versus DOST in female wearing high heels and its impact on posture.

DETAILED DESCRIPTION:
The consequences of wearing high heels included increased bending of the hips and knees, anterior pelvic tilting, and increased lumbar lordosis in the spine. Wearers of high heels reported reduced dorsiflexion. The aim of this study is to compare the effectiveness of Graston technique and Dynamic Oscillatory Stretch (DOST) technique in improving lumbar lordosis, anterior pelvic tilting and function status in high heel users. This study is randamized control trial. The sample size of this study is 30 participants which would be divided into two group, 15 each. Non-probability Convenience sampling will be used and participants are randomly assigned into Group A (Graston Technique) Group B (DOST) through envelope sealed method after baseline assessment . The participants of both group were evaluated on three occasions; (i) baseline, (ii) 5th session and (iii) 12th session.

ELIGIBILITY:
Inclusion Criteria:

* • Only female were included

  * Age group 20 to 40 years.
  * Duration of wearing HH: >1 yr.
  * Wearing HH for > 3 times a wk. and 5 hrs/ day.
  * Heel height: 2 inch and above
  * Decreased ankle Dorsiflexion (less than 17 degrees)
  * Lumber lordosis increased (> 40).
  * Muscle tightness (Paraspinal, hamstring, gastrocnemius and soleus).

Exclusion Criteria:

* • DVT, malignancy, infection.

  * Eczema or other skin diseases.
  * MSK injury or surgery of LL.
  * Sciatica or other Neuropathy/ Neurological disorder
  * Acute Cardio-Respiratory disorder

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 30 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Flexicurve Ruler | 3 week
  The Flexicurve ruler allows us to measure the curves of your spine. The Flexicurve is a strip of flexible metal covered in plastic. It will place at the top of the back then gently bend it so it reflects the shape of the backbone.
Inclinometer | 3 week
  Inclinometer is a specialized tool used to measure angles and range of motion of joints. It is used to measure pelvic tilt.

SECONDARY OUTCOMES:
Gonimeter | 3 week
  A device that measures an angle or allows an object to be rotated to a certain position. In orthopedics, the former description is more accurate. Goniometry is the art and science of measuring joint ranges in each plane of the joint
Lower Extremity Functional Scale | 3 week
  The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, Principal Investigator — Riphah International University
Locations (1):
- Gulberg Green Campus of Riphah International University, Islamabad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien HL, Lu TW, Liu MW. Effects of long-term wearing of high-heeled shoes on the control of the body's center of mass motion in relation to the center of pressure during walking. Gait Posture. 2014 Apr;39(4):1045-50. doi: 10.1016/j.gaitpost.2014.01.007. Epub 2014 Jan 19. PMID 24508016